CLINICAL TRIAL: NCT04297241
Title: Nitrate Effect on Exercise Capacitance and Hemodynamic Profile Prior to Fontan Failure
Brief Title: Nitrate Effect on Exercise Capacitance
Acronym: NEET
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018-0020
Record Dates: First submitted 2020-02-05; First posted 2020-03-05 (Actual); Results first posted 2021-08-25 (Actual); Last update posted 2021-09-22 (Actual); Status verified 2021-07

CONDITIONS: Fontan
MeSH Terms: interventions — Isosorbide Dinitrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Isosorbide Dinitrate (Experimental): Each enrolled participant will be on a titrated dosage of isosorbide dinitrate to determine effectiveness on both primary and secondary outcome measures.
  Interventions: Drug: Isosorbide Dinitrate

INTERVENTIONS:
Drug: Isosorbide Dinitrate — All patients will be given a 6 week titration regimen of study medication. Patients will begin at a 5mg dosage and titrate up to 30mg three times per day if each subsequent dose is tolerated.
  Other Names: Isordil

SUMMARY:
The investigators will investigate the safety and preliminary efficacy of ISDN therapy to reduce venous congestion and improve exercise tolerance in children and adults after the Fontan operation. This will be accomplished by recruiting 15 Fontan physiology patients from the Cincinnati Children's Fontan clinic and University of Kentucky Pediatric Cardiology clinic for the investigation. The investigators will non-invasively measure both central venous pressures at rest and during graded cardiopulmonary exercise testing. In addition the study team will obtain a measurement of liver stiffness before and after a 4-week regimen of ISDN therapy. Patients will be seen twice in clinic, once before and after ISDN therapy, and phone calls will be made to ensure safety, compliance, and make appropriate alterations to medications throughout the study period. Pre- and post-intervention central venous pressure and exercise tolerance will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Underlying Fontan physiology
* On a stable medication regimen for the past 3 months
* Nine years of age or older

Exclusion Criteria:

* Pregnant or nursing
* Prior hospitalization for heart failure in past year
* Presence of uncontrolled arrhythmias within the past 6 months
* Non-cardiac conditions which significantly limited exercise
* Moderate or severe ventricular dysfunction by echocardiogram or cardiac MRI
* Currently treated with a phosphodiesterase-5 inhibitor or organic nitrates
* Concurrent enrollment in other investigational drug trial
* End stage Liver Disease (ESLD)

Min Age: 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-12-12 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2021-05-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Cincinnati Childrens Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bigelow AM, Riggs KW, Morales DLS, Opotowsky AR, Lubert AM, Dillman JR, Veldtman GR, Heydarian HC, Trout AT, Cooper DS, Goldstein SL, Chin C, Palermo JJ, Ollberding NJ, Mays WA, Alsaied T. Isosorbide DiNitrate Effect on Hemodynamic Profile, Liver Stiffness, and Exercise Tolerance in Fontan Circulation (The NEET Clinical Trial). Pediatr Cardiol. 2024 Oct;45(7):1389-1397. doi: 10.1007/s00246-023-03156-3. Epub 2023 Apr 21. PMID 37084132

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a prospective study to evaluate the safety and efficacy of isosorbide dinitrate in children and adults with Fontan physiology in decreasing liver stiffness and lowering exercise related venous pressure responses and increasing exercise tolerance who are ≥ 9 years old. Each patient completed a total of 6 study visits over the course of 2 years.
Pre-assignment Details: Each patient came in for a baseline assessment visit. At the end of the baseline visit, they received isosorbide dinitrate, which began at a small dose (5 mg three times daily) and were titrated up to three times daily over 2 weeks. The medication was continued for 4 weeks once the target dose was reached. At the end of 4 weeks, the participants returned for a final visit.
Groups:
- Isosorbide Dinitrate: All patients will have a baseline assessment immediately preceding initiation of isosorbide dinitrate. This will include vitals, urine pregnancy test for all females, blood collection, insertion of a peripheral venous cannula for venous blood pressure during exercise testing, maximal cardiopulmonary exercise testing/Ramp protocol including spirometry, and liver ultrasound to assess for liver stiffness.
  All patients will then be given a 6 week titration regimen of study medication. Patients will begin at a 5mg dosage and titrate up to 30mg three times per day if each subsequent dose is tolerated.
  Four follow-up phone calls will take place every 3 days to ensure the patient is tolerating the medication and a medication adjustment will occur as needed.
  Approximately 4 weeks after study drug administration, participants will return for the same tests/procedures as performed during the baseline visit.
Period: Overall Study
Arm/Group | Isosorbide Dinitrate
Started | 20
Completed | 15
Not Completed | 5
Not completed — Withdrawal by Subject | 1
Not completed — Adverse Event | 1
Not completed — Physician Decision | 3

BASELINE CHARACTERISTICS:
Groups:
- Isosorbide Dinitrate: Isosorbide Dinitrate: This is a prospective study in children and adults with Fontan physiology to see if isosorbide dinitrate will be safely tolerated and improve exercise venous pressure responses, as well as exercise tolerance in Fontan patients. Participants will receive isosorbide dinitrate as a small dose (5 mg three times daily) and titrate up to three times daily over 2 weeks. The medication will continue for 4 weeks once the target dose is reached.
Arm/Group | Isosorbide Dinitrate
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 5
  Between 18 and 65 years | 15
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 18
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experience an Adverse Reaction to the Study Medication During the Study Enrollment Period.
Description: Potential adverse side effects of study medication (isosorbide dinitrate) will be monitored throughout study period. Study medication will be titrated to a maximal dose of 30mg dependent on the patient tolerance. Patient tolerance is defined by frequency of known risk factors to the study medication (headaches, hypotension, and syncope).
Time Frame: Baseline and 6 weeks
Population: Adverse Events
Measure: Count of Participants; unit: Participants
Groups:
- Isosorbide Dinitrate: Determine the number of participants who experience an adverse reaction to the study medication during the study enrollment period.
Arm/Group | Isosorbide Dinitrate
Number analyzed (Participants) | 20
Participants | 16

2. Secondary Outcome: Effect of Isosorbide Dinitrate on Liver Stiffness Levels
Description: Determine effectiveness of study medication on hemodynamic profile by completing baseline and post-study medication liver ultrasound measuring liver stiffness levels by sheer wave speed (m/s).
Time Frame: Baseline and 6 weeks
Population: Hemodynamic profile
Measure: Median (Standard Deviation); unit: m/s
Groups:
- Isosorbide Dinitrate - Baseline; Isosorbide Dinitrate - Post-therapy: Determine effectiveness of study medication on hemodynamic profile by completing baseline and post-study medication liver ultrasound measuring liver stiffness levels.
Arm/Group | Isosorbide Dinitrate - Baseline | Isosorbide Dinitrate - Post-therapy
Number analyzed (Participants) | 20 | 20
m/s | 2.3 (0.4) | 2.1 (0.5)

3. Secondary Outcome: Effect of Isosorbide Dinitrate on Central Venous Pressure
Description: Determine effectiveness of study medication on hemodynamic profile by completing baseline and post-study medication maximal exercise tests to measure central venous pressure via IV catheter insertion
Time Frame: Baseline and 6 weeks
Measure: Median (Standard Deviation); unit: mmHg
Groups:
- Isosorbide Dinitrate - Baseline; Isosorbide Dinitrate - Post-therapy: Determine effectiveness of study medication on hemodynamic profile by completing baseline and post-study medication maximal exercise tests to measure central venous pressure via IV catheter insertion
Arm/Group | Isosorbide Dinitrate - Baseline | Isosorbide Dinitrate - Post-therapy
Number analyzed (Participants) | 20 | 20
mmHg | 22.5 (4.5) | 20.6 (2.9)

4. Secondary Outcome: Effect of Isosorbide Dinitrate on Maximal Exercise Capacity VO2 Max
Description: Obtain estimates of the effect the study medication has on maximal exercise test VO2 max performance in Fontan patients by study participants performing a maximal ramp exercise test on a stationary bike.
Time Frame: Baseline and 6 weeks
Measure: Median (Standard Deviation); unit: mL/min
Groups:
- Isosorbide Dinitrate - Baseline; Isosorbide Dinitrate - Post-therapy: Obtain estimates of the effect the study medication has on maximal exercise test VO2 max performance in Fontan patients by study participants performing a maximal ramp exercise test on a stationary bike.
Arm/Group | Isosorbide Dinitrate - Baseline | Isosorbide Dinitrate - Post-therapy
Number analyzed (Participants) | 20 | 20
mL/min | 1086.7 (312.9) | 1151.3 (301.5)

5. Secondary Outcome: Effect of Isosorbide Dinitrate on Maximal Exercise Capacity Heart Rate Response
Description: Obtain estimates of the effect the study medication has on maximal exercise test heart rate response in Fontan patients by study participants performing a maximal ramp exercise test on a stationary bike.
Time Frame: Baseline and 6 weeks
Measure: Median (Standard Deviation); unit: bpm
Groups:
- Isosorbide Dinitrate - Baseline; Isosorbide Dinitrate - Post-therapy: Obtain estimates of the effect the study medication has on maximal exercise test heart rate response in Fontan patients by study participants performing a maximal ramp exercise test on a stationary bike.
Arm/Group | Isosorbide Dinitrate - Baseline | Isosorbide Dinitrate - Post-therapy
Number analyzed (Participants) | 20 | 20
bpm | 156.6 (26.4) | 164.7 (22.1)

6. Secondary Outcome: Effect of Isosorbide Dinitrate on Maximal Exercise Capacity Respiratory Rate Response
Description: Obtain estimates of the effect the study medication has on maximal exercise test respiratory rate response in Fontan patients by study participants performing a maximal ramp exercise test on a stationary bike.
Time Frame: Baseline and 6 weeks
Measure: Median (Standard Deviation); unit: Respiratory Exchange Ratio
Groups:
- Isosorbide Dinitrate - Baseline; Isosorbide Dinitrate - Post-therapy: Obtain estimates of the effect the study medication has on maximal exercise test respiratory rate response in Fontan patients by study participants performing a maximal ramp exercise test on a stationary bike.
Arm/Group | Isosorbide Dinitrate - Baseline | Isosorbide Dinitrate - Post-therapy
Number analyzed (Participants) | 20 | 20
Respiratory Exchange Ratio | 1.17 (0.09) | 1.19 (0.09)

ADVERSE EVENTS:
Time Frame: Isosorbide Dinitrate therapy was initiated at a low dose (e.g. 5 mg three times daily in patients above 50 kg) and increased incrementally over 2 weeks to a goal of 30 mg three times a day. The medication was then continued for approximately 4 weeks once the target dose was achieved for a total of 6 weeks.
Groups:
- Isosorbide Dinitrate: Isosorbide Dinitrate therapy was initiated at a low dose (e.g. 5 mg three times daily in patients above 50 kg) and increased incrementally over 2 weeks to a goal of 30 mg three times a day. The medication was then continued for approximately 4 weeks once the target dose was achieved for a total of 6 weeks.
Arm/Group | Isosorbide Dinitrate
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 1/20
Other Adverse Events (participants affected / at risk) | 16/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Isosorbide Dinitrate (N=20)
Study Medication Overdose (Cardiac disorders) | 1 (1) — Patient understanding of medication dosage calendar was not correct upon completion of initial study visit, therefore patient took a higher dose of medication at the beginning of study participation and needed to restart the study.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Isosorbide Dinitrate (N=20)
Headache (Nervous system disorders) | 16 (23)
Fluttering (Cardiac disorders) | 1 (1)
Skipped heart beat (Cardiac disorders) | 1 (1)
Sinus infection (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dizziness (Nervous system disorders) | 2 (2)
Tachycardia (Cardiac disorders) | 2 (2)
Jittery (Nervous system disorders) | 1 (1)
Agitation (Nervous system disorders) | 1 (1)
Arm pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Lightheaded (Vascular disorders) | 2 (2)
Burning chest (Cardiac disorders) | 1 (2)
Pain in extremities (Musculoskeletal and connective tissue disorders) | 1 (1)
Tingling in extremities (Musculoskeletal and connective tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-12-16): https://cdn.clinicaltrials.gov/large-docs/41/NCT04297241/Prot_SAP_000.pdf